CLINICAL TRIAL: NCT00003892
Title: Phase II Study of CGP 69846A (ISIS 5132) in Recurrent Epithelial Ovarian Cancer
Brief Title: ISIS 5132 in Treating Patients With Metastatic or Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I116; CAN-NCIC-IND116 (Other: PDQ); CDR0000067061 (Other: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-08-05 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Ovarian Cancer
Keywords: stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — ISIS 5132

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ISIS 5132 (Experimental): ISIS 5132 x 21 days IV infusion
  Interventions: Drug: ISIS 5132

INTERVENTIONS:
Drug: ISIS 5132 — 4mg/kg/day IV for 21 days every 4 weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of ISIS 5132 in treating patients who have metastatic or recurrent ovarian cancer that has not responded to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of ISIS 5132 by evaluating objective response and duration of response in patients with recurrent ovarian epithelial cancer. II. Determine the tolerability and quantitative toxicity of ISIS 5132 in this patient population.

OUTLINE: This is a multicenter study. Patients receive ISIS 5132 IV continuously for 21 days. Courses are repeated every 28 days. Treatment continues for a maximum of 12 courses in the absence of disease progression or unacceptable toxicity. Patients with documented complete response receive an additional 2 courses. Patients with documented partial response receive an additional 4 courses. Patients are followed at 4 weeks, then every 3 months until disease relapse or progression.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study over 12-15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically documented ovarian epithelial cancer Metastatic and/or locally recurrent disease that is incurable with standard therapy Must have received 1 or 2 prior regimens of chemotherapy At least 1 regimen must have contained cisplatin or carboplatin Bidimensionally measurable disease Indicator lesion size must be as follows: At least 4-50 cm2 by CT scan At least 1 cm2 by chest xray At least 1 cm2 (e.g., nodules) by physical exam No abdominal adenocarcinoma of unknown origin No borderline ovarian tumor No tumor known to be of primary fallopian tube or peritoneal origin

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: At least 12 weeks Hematopoietic: Platelet count at least 100,000/mm3 Absolute granulocyte count at least 1,500/mm3 No known bleeding disorder Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) AST less than 5 times ULN PT/PTT normal (except when elevated due to therapeutic coumadin) Renal: Creatinine no greater than 2 times ULN Cardiovascular: No significant cardiac dysfunction Neurologic No history of significant neurologic disorder No significant psychiatric disorder Other: Not pregnant or nursing Fertile patients must use effective contraception At least 5 years since prior malignancy and no evidence of recurrence No other serious illness or medical condition No active uncontrolled infection No complete bowel obstruction

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy No other concurrent cytotoxic therapy Endocrine therapy: Not specified Radiotherapy: Recovered from prior radiotherapy At least 4 weeks since radiotherapy to at least 20% of bone marrow Surgery: Not specified Other: As least 28 days since prior investigational agent or new anticancer therapy No concurrent therapeutic heparin No other concurrent investigational therapy

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 1999-02-01 (Actual); Primary Completion 2000-10-17 (Actual); Study Completion 2008-09-22 (Actual)

PRIMARY OUTCOMES:
Objective and duration of response | 9 years
  To determine the efficacy of ISIS 5132 in patients with recurrent epithelial ovarian cancer, with evaluation of objective responses and duration of responses in patients receiving this compound in a phase II trial.

SECONDARY OUTCOMES:
Toxicity | 9 years
  To determine the tolerability and quantitative toxicity of ISIS 5132 when given to patients with recurrent ovarian cancer

CONTACTS AND LOCATIONS:
Overall Officials: Amit M. Oza, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (66):
- United States (2):
  - Duluth Clinic, Duluth, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
- Canada (63):
  - Cross Cancer Institute, Edmonton, Alberta
  - Lethbridge Cancer Clinic, Lethbridge, Alberta
  - Burnaby Hospital Regional Cancer Centre, Burnaby, British Columbia
  - Penticton Regional Hospital, Penticton, British Columbia
  - British Columbia Cancer Agency - Fraser Valley Cancer Centre, Surrey, British Columbia
  - Prostate Centre at Vancouver General Hospital, Vancouver, British Columbia
  - BC Cancer Agency, Vancouver, British Columbia
  - St. Paul's Hospital - Vancouver, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Queen Elizabeth II Health Science Center, Halifax, Nova Scotia
  - Royal Victoria Hospital, Barrie, Barrie, Ontario
  - Peel Memorial Hospital, Brampton, Ontario
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - York County Hospital, Newmarket, Ontario
  - North York General Hospital, Ontario, North York, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Regional Cancer Center - General Division, Ottawa, Ontario
  - Ottawa Regional Cancer Centre - Civic Campus, Ottawa, Ontario
  - Peterborough Oncology Clinic, Peterborough, Ontario
  - Algoma District Medical Group, Sault Ste. Marie, Ontario
  - Scarborough Hospital - General Site, Scarborough Village, Ontario
  - Hotel Dieu Hospital - St. Catharines, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Women's College Campus, Sunnybrook and Women's College Health Science Center, Toronto, Ontario
  - Saint Joseph's Health Centre - Toronto, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - Queen Elizabeth Hospital, PEI, Charlottetown, Prince Edward Island
  - Centre Universitaire de Sante de l'Estrie, Fleurimont, Quebec
  - Centre Hospitalier Regional de Lanaudiere, Joliette, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - Hotel Dieu de Montreal, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Centre Hospitalier de l'Universite' de Montreal - Pavillon Saint-Luc, Montreal, Montreal, Quebec
  - Royal Victoria Hospital - Montreal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec
  - Queen Elizabeth Hospital, Montreal, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Pavillion de Quebec, Québec, Quebec
  - Hopital du Saint-Sacrament, Quebec, Québec, Quebec
  - Hopital du Haut-Richelieu, Saint-Jean-sur-Richelieu, Quebec
  - Hopital Laval, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Royal South Hants Hospital, Southampton, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oza AM, Elit L, Swenerton K, Faught W, Ghatage P, Carey M, McIntosh L, Dorr A, Holmlund JT, Eisenhauer E; NCIC Clinical Trials Group Study (NCIC IND.116). Phase II study of CGP 69846A (ISIS 5132) in recurrent epithelial ovarian cancer: an NCIC clinical trials group study (NCIC IND.116). Gynecol Oncol. 2003 Apr;89(1):129-33. doi: 10.1016/s0090-8258(02)00144-0. PMID 12694666